CLINICAL TRIAL: NCT05052346
Title: Association of the Neutrophil/Lymphocyte Ratio and Lymphocyte/Platelet Ratio With Pulmonary Complications and Mortality in COVID-19 Patients
Brief Title: Association of the Neutrophil/Lymphocyte Ratio With Pulmonary Complications and Mortality in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Christian Omar Ramos-Peñafiel, MD, PhD, Principal Investigator, Hospital General de Mexico
Other Study IDs: NR-09-2020
Record Dates: First submitted 2020-07-31; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Pulmonary Complication
Keywords: Pulmonary Complications; Mortality; COVID-19; Neutrophil/Lymphocyte Ratio
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Coronavirus Disease-19 (COVID-19) pandemic is currently a priority for health services worldwide. Unlike the Severe Acute Respiratory Syndrome-Coronavirus (SARS-CoV) epidemic in 2012, the COVID-19 shows specific alterations in the white blood cell count, accentuated in severe cases, and with respiratory failure. Among the most relevant data are both lymphopenia, thrombocytopenia, and eosinopenia. The Neutrophil Lymphocyte Index has been beneficial in the evaluation of infectious respiratory processes, showing a sensitivity similar to scales such as CURB65 (Confusion, Uremia, Respiratory rate, BP, age ≥ 65 years). Because COVID-19 infection shows alterations in the blood cell ratio, these indices may be useful in evaluating patients with COVID-19 infection.

DETAILED DESCRIPTION:
The hematological alterations in patients with COVID-19 divided into two aspects: the main ones, the global leukocyte count, and the individual counts. Most of the information about the behavior of blood counts come from cases attended in Wuhan, China. At the Zhongnan Hospital in Hubei Province, identified that the lymphocyte count was lower in critically ill patients. At the same time, the leukocyte counts were higher in deaths associated with COVID-19, this elevation being mainly of neutrophils. The lymphopenia is also a constant data in COVID-19 (47.4%), especially in cases that entered the Intensive Care Unit. As in community pneumonia, severe lymphopenia has associated with a high risk of death. A relationship between neutrophils and lymphocytes is called the Neutrophil-Lymphocyte index. This index is especially useful for predicting respiratory complications, such as for COVID-19, where mortality ranges from 2-9% compared to the 2012 epidemic (10%) or Middle East Respiratory Syndrome (37%). In Mexico, there is a high prevalence of chronic diseases that increase the risk of COVID-19 infection. This study's main objective is to identify the association of blood abnormalities on respiratory complications associated with COVID-19 infection. All data were obtained from the clinical records of patients treated by COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active COVID-19 infection

Exclusion Criteria:

* Liver failure
* Active cancer
* Chronic renal failure
* AIDS
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican patients diagnosed with active COVID-19 infection who require hospital care and who have peripheral blood counts at diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Respiratory Complications in COVID-19 patients | 6 months
  To assess the relationship of the Neutrophil-Lymphocyte and Lymphocyte-Platelet index on respiratory complications
Mortality in COVID-19 patients | 6 months
  To assess the relationship of the Neutrophil-Lymphocyte and Lymphocyte-Platelet index on respiratory complications

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Martinez Tovar, Study Director — Hospital General de Mexico
Locations (1):
- Omar Ramos-Peñafiel, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
All participants and their information will be managed by intern investigators and will be kept secure for personal data protection according to Mexican laws